CLINICAL TRIAL: NCT05572502
Title: The Feasibility, Implementation and Efficacy of a Diabetes Reversal Online Program and Study (DROP Study) in an Office Setting
Brief Title: Diabetes Reversal Online Program and Study (DROP Study)
Acronym: DROP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Principal Investigator, Vanita Rahman, Clinic Director, Physicians Committee for Responsible Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00066361
Record Dates: First submitted 2022-10-03; First posted 2022-10-07 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
Keywords: plant-based; vegan; diet; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Diet, Plant-Based; Diet, Vegan

STUDY DESIGN:
Intervention Model Description: single group, multiple replications
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vegan diet (Experimental): All participants will follow a low-fat vegan diet. There are no other study arms or control group.
  Interventions: Behavioral: plant-based diet

INTERVENTIONS:
Behavioral: plant-based diet — For the duration of the study, this arm will: follow a low-fat vegan diet; weigh themselves weekly, and get fasting bloodwork before, during and after the study
  Other Names: vegan diet

SUMMARY:
This is an interventional study that will evaluate the feasibility, implementation, and efficacy of an online, 12-week, plant-based, nutrition education program in a community setting. Data will also be analyzed to see if participation in the program results in reductions glycated hemoglobin levels, body weight, and cholesterol levels.

DETAILED DESCRIPTION:
This study aims to assess the feasibility and implementation of an online, plant-based, diabetes reversal program in a community setting. The study will also assess changes in glycated hemoglobin, body weight, and plasma lipids with an online 12-week, plant-based, nutrition education program. These health benefits may illustrate feasibility to physicians and healthcare professionals elsewhere, in addition to their value for the individual research participants.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Men and women meeting the age of majority, defined as follows: Age 19 or older in Nebraska and Alabama; Age 21 or older in Mississippi; Age 18 or older in all other states
* Prior diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

* Use of recreational drugs in the past 6 months
* Pregnancy or intention to become pregnant during the study period, as verified by self-report
* Unstable medical or psychiatric illness
* Lack of English fluency
* Inability to maintain current medication regimen
* Inability or unwillingness to participate in all components of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-08-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 12 weeks
  A1c will be measured before and after the study period

SECONDARY OUTCOMES:
body weight | 12 weeks
  participants will track body weight weekly using a RNFO scale
total cholesterol | 12 weeks
  total cholesterol will be measured before and after the study period
LDL cholesterol | 12 weeks
  LDL cholesterol will be measured before and after the study period
medication usage | 12 weeks
  changes in medications to treat diabetes will be tracked during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physician Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tonstad S, Butler T, Yan R, Fraser GE. Type of vegetarian diet, body weight, and prevalence of type 2 diabetes. Diabetes Care. 2009 May;32(5):791-6. doi: 10.2337/dc08-1886. Epub 2009 Apr 7. PMID 19351712
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Background] Barnard N, Scherwitz L, Ornish D. Adherence and acceptability of a lowfat vegetarian diet among patients with cardiac disease. J Cardiopulmonary Rehabil 1992;12:423-31.
- [Background] Barnard N, Scialli A, Bertron P, Hurlock D, Edmonds K. Acceptability of a therapeutic low-fat, vegan diet in premenopausal women. J Nutr Educ 2000;32:314-9.
- [Background] Barnard ND, Scialli AR, Turner-McGrievy G, Lanou AJ. Acceptability of a low-fat vegan diet compares favorably to a step II diet in a randomized, controlled trial. J Cardiopulm Rehabil. 2004 Jul-Aug;24(4):229-35. doi: 10.1097/00008483-200407000-00004. PMID 15286527
- [Background] Barnard ND, Gloede L, Cohen J, Jenkins DJ, Turner-McGrievy G, Green AA, Ferdowsian H. A low-fat vegan diet elicits greater macronutrient changes, but is comparable in adherence and acceptability, compared with a more conventional diabetes diet among individuals with type 2 diabetes. J Am Diet Assoc. 2009 Feb;109(2):263-72. doi: 10.1016/j.jada.2008.10.049. PMID 19167953
- [Background] American Dietetic Association; Dietitians of Canada. Position of the American Dietetic Association and Dietitians of Canada: Vegetarian diets. J Am Diet Assoc. 2003 Jun;103(6):748-65. doi: 10.1053/jada.2003.50142. PMID 12778049
- [Background] Barnard ND, Akhtar A, Nicholson A. Factors that facilitate compliance to lower fat intake. Arch Fam Med. 1995 Feb;4(2):153-8. doi: 10.1001/archfami.4.2.153. PMID 7842153
- [Background] Becker M. The health belief model and personal health behavior. Health Education Monographs 1974;2:324-473.
- [Background] U.S. Census Bureau. Quick Facts. Internet: https://www.census.gov/quickfacts/fact/table/US/PST045221, accessed July 5, 2022.